CLINICAL TRIAL: NCT02297750
Title: Optimal Timing of Double-Wire Technique For Biliary Cannulation at ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00033706
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2014-11

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: The focus of the study is double-wire technique versus single wire technique in patients undergoing ERCP with biliary cannulation as the primary objective.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single wire technique (Active Comparator): single wire technique in patients undergoing ERCP with biliary cannulation
  Interventions: Procedure: single-wire technique in patients undergoing ERCP with biliary cannulation
- Double wire technique (Active Comparator): double-wire technique in patients undergoing ERCP with biliary cannulation
  Interventions: Procedure: double-wire technique in patients undergoing ERCP with biliary cannulation

INTERVENTIONS:
Procedure: double-wire technique in patients undergoing ERCP with biliary cannulation
  Arms: Double wire technique
Procedure: single-wire technique in patients undergoing ERCP with biliary cannulation
  Arms: single wire technique

SUMMARY:
The purpose of this study is to give doctors who perform Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures a better idea as to the best techniques to use in order to examine the bile duct as quickly and safely as possible.

DETAILED DESCRIPTION:
Sometimes, in the course of a regular ERCP procedure, techniques used by the doctor to pass a wire into the bile duct can result in the pancreas duct being entered instead. When this happens, the doctor may either remove the wire (known as "single wire" technique) or leave it in and use a second wire ("double wire") to enter the bile duct. This study will try to determine whether the "double wire" technique or the "single wire" technique removing the wire is the safest and most efficient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ERCP with primary intent to cannulate the bile duct
2. Written informed consent

Exclusion Criteria:

1. Age < 18 years
2. Non-naive papilla (previous sphincterotomy)
3. Surgically altered anatomy
4. Known/suspected pancreas divisum
5. Suspected SOD/biliary manometry
6. Prior ERCP/stent within 3 months
7. ERCP performed in the Operating Room or at Duke North
8. Pregnancy/breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Success of biliary cannulation | 10 minutes after randomization
  The primary outcome is incidence of successful deep biliary cannulation within 10 minutes.

SECONDARY OUTCOMES:
Success of biliary cannulation | 2 days after the procedure
  Number of attempts required for successful biliary cannulation
Time to successful biliary cannulation | 2 days after the procedure
Post-ERCP pancreatitis | 2 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mahfuzul Haque, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States